CLINICAL TRIAL: NCT04216992
Title: Institutional Review Board of Tri-Service General Hospital, National Defense Medical Center
Brief Title: Value of Three-dimensional Rotational Epidurography on Percutaneous Epidural Adhesiolysis
Status: Completed | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, yi-chih HSU, Assistant professor, Tri-Service General Hospital
Other Study IDs: 1-105-05-141
Record Dates: First submitted 2019-12-28; First posted 2020-01-03 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Failed Back Surgery Syndrome; Spinal Stenosis
Keywords: Cone beam; Computed tomography; Epidurography; Percutaneous epidural adhesiolysis
MeSH Terms: conditions — Failed Back Surgery Syndrome; Spinal Stenosis | interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Three dimensional-rotational epidurography (3D-RE): 3D-RE is obtained on a commercial digital bi-plane angiography system. Reconstruction time was 30 seconds. Detailed information regarding technical performance and reconstruction procedure has been reported. Postprocessing techniques provided by the software included real-time 3D volume rendering and multiplanar reformatting. Real-time 3D volume rendering creates a 3D model of the examined object. The software allows emphasizing bony structures or soft tissue by changing intensity, brightness, and opacity of different X-ray structures. Additionally, rotation of the 3D object in all directions is possible, as is a virtual stereoscopic view provided by the software in combination with special glasses. The multiplanar reformatting modus generates virtual sections according to the three main axes and free defined axes. The section planes can be freely chosen, and curved sectioning is also possible.
  Interventions: Device: Cone beam computed tomography

INTERVENTIONS:
Device: Cone beam computed tomography — The contrast agent (Omnipaque, GE Healthcare, Ireland) was instilled to conﬁrm the epidural space. With use of a calibrated angiographic C-arm system and a postprocessing workstation, we acquired volume data sets from two dimensional digital projection images obtained to reconstruct the 3D-RE during a C-arm rotation around the patient axis.

SUMMARY:
Conventional epidurography (CE) is thought to have insufficient usefulness on percutaneous epidural adhesiolysis (PEA). The investigators aimed to evaluate the association between the outcome of PEA and three dimensional-rotational epidurography (3D-RE). The investigators performed 30 PEA in 26 patients, and evaluated their post-PEA image findings. Two independent clinicians categorized and recorded the occurrence of contrast at intra-canal ventral and extra-foraminal regions on CE; and contrast at dorsal canal (DC), ventral canal (VC), dorsal foramen (DF), and ventral foramen (VF) on 3D-RE. Reproducibility was assessed using intra-class correlation coefficients (ICCs). The symptom relief after one month for the patients receiving PEA and the contrast distribution patterns of CE and 3D-RE and were determined.

DETAILED DESCRIPTION:
Patient Selection. This prospective study protocol was approved by the ethics committee, and informed consent was obtained from all subjects. The investigators analyzed the medical and radiographic records included patients who underwent lumbar PEA procedures at a single university hospital. The inclusion criterion was FBSS and SS with unilateral radiculopathy. All patients reported a history of discogenic or radicular symptoms refractory to conservative treatments and epidural steroid injection for a minimum of 6 weeks. Diagnoses were established using magnetic resonance imaging (MRI) and/or computed tomography (CT) performed before PEA. The PEA was standardized to all patients receiving the procedure. Each patient received an epidural injection, and if the symptoms persisted or the relief was insufficient, the patient received PEA >6-week interval between the epidural steroid injection. Positive provocative test during PEA was used to confirm the affected spinal level [11]. All patients underwent CE before and after PEA; and 3D-RE after PEA. Patients with a history of spinal surgery and those with cauda equina syndrome, bleeding diathesis, associated somatic or psychiatric disease, vertebral fractures, pregnancy, and tumors or other underlying systemic diseases that could signiﬁcantly aﬀect the procedural outcomes were excluded. The patients had bilateral symptoms and did not react to the provocation during PEA were also excluded. All procedures were performed by one of the authors (YCH) using the same procedural protocol.

PEA Procedure. A standard PEA procedure was used to lyse adhesions and achieve nerve blockades in all patients, as previously described [1,2]. A 1-day standardized protocol was followed. The patient was placed on a radiolucent table in the prone position, and the procedure was performed under ﬂuoroscopic guidance. The coccygeal and sacral regions were disinfected with 10% Betadine, and the surgical site was draped in the usual aseptic manner. The sacral hiatus was anesthetized with 1% xylocaine. Then, a 13.6-G Coaxial needle was introduced into the epidural space below the level of S3 with a combined use of US-guidance and fluoroscopy insurance. The US was provided using a scanner (Xario 100; Toshiba, Tokyo, Japan) with a 7~18 MHz linear transducer (PLU-1204BT). A total of 0.5 mL of the contrast agent (Omnipaque, GE Healthcare, Ireland) was instilled to conﬁrm the epidural space. Both anteroposterior, right-oblique, left-oblique, and lateral ﬂuoroscopic views were obtained. The investigators also assessed the development of any adverse reactions. On conﬁrmation of the target for PEA, an angiographic catheter (Cobra 4-Fr; Cordis, USA) and/or coaxial supporting catheter (Chiba 6-Fr; Cook, USA) was gently inserted toward the target site. Once it reached the target site, a second CE was obtained by injecting 3 mL of the contrast agent for the identiﬁcation of ﬁlling defects or cutoﬀ signs surrounding the target area. The investigators choose the target nerve roots for PEA by clinical dermatome involvement and provocation tests during PEA. The catheter tip was positioned at the ventral epidural space of the target site, and in the case of foraminal diseases, was placed at the opening of the foramen [12]. When the tip of the catheter touched the target site or the contrast agent exerted pressure on the lesion, patients were asked to report provoked symptoms [4]. According to the surgical records, they frequently reported pain similar to what they had been suﬀering. Both mechanical and fluid adhesiolysis were performed. The former was achieved through pushing, pulling, and rotating movements of the catheter, while the latter was achieved by the injection of 0.9% normal saline (10 mL). Following PEA, a third CE and 3D-RE was obtained using 3 mL of the contrast agent. All CE and 3D-RE images were saved in the Digital Imaging and Communications in Medicine format for future analysis, and the CE and 3D-RE after PEA was used for analysis in our study. Finally, a 40 mg triamcinolone acetonide (YungShin, Taichung, Republic of China) was slowly injected.

3D-RE technique. After performing PEA, 3D-RE are obtained on a commercial digital bi-plane angiography system (Allura Xper, Philips). A 240-degree rotation forward and backward of the tube-camera unit around the patient's longitudinal axis within 4 seconds is performed by using an acquisition matrix of 1024 x 1024 pixels. The forth and back rotation results in 120 radiographs. Raw data were automatically sent to a dedicated workstation (Philips Xtra vision workstation), where the rotational projection images are prepared for computed 3D reconstruction. 2D radiographs are used to determine the volume of interest. After correction of gain and distortion, a 3D data set is calculated, resulting in 512 transverse CT-equivalent sections. Depending on the initially chosen volume of interest, the voxel size varies from 0.1 to 0.6 mm. The investigators used a resolution of 0.14-mm voxel size, which resulted in a 3D cuboid of 25 x 19 x 25 cm.

Reconstruction time was 30 seconds. Detailed information regarding technical performance and reconstruction procedure has been reported [13]. Postprocessing techniques provided by the software included real-time 3D volume rendering and multiplanar reformatting. Real-time 3D volume rendering creates a 3D model of the examined object. The software allows emphasizing bony structures or soft tissue by changing intensity, brightness, and opacity of different X-ray structures. Additionally, rotation of the 3D object in all directions is possible, as is a virtual stereoscopic view provided by the software in combination with special glasses. The multiplanar reformatting modus generates virtual sections according to the three main axes and free defined axes. The section planes can be freely chosen, and curved sectioning is also possible.

Conventional epidurography and 3D-RE Contrast Distributions. Post-PEA CE contrast patterns were deﬁned and classiﬁed into 2 types according to the system proposed by Park et al. and Gupta et al.[4,6]: Limited intracanal ventral spread (ICV) and extended extraforaminal spread (EF) (Figure 1). The investigators defined the contrast distributions into 4 areas by post-PEA 3D-RE : Dorsal Canal (DC), contrast spread to the dorsal zone of the ipsilateral epidural space not extending to the neural foramen; Ventral Canal (VC), contrast spread to the ventral zone of the ipsilateral epidural space not extending to the neural foramen; Dorsal Foramen (DF), contrast spread to the dorsal zone of the ipsilateral epidural space extending to the neural foramen; Ventral Foramen (VF), contrast spread to the ventral zone of the ipsilateral epidural space extending to the neural foramen (Figure 2). The CE and 3D-RE images were analyzed and recorded by a musculoskeletal radiologist (Y.C.H.) and a surgeon (C.T.T.) who blinded to the results of the clinical data. The investigators made a consensus if there was discrepancy between the analyses of these images.

Data collection. All patients were clinically evaluated before and 1 month after PEA by a nurse specialized in pain management and blinded to the treatment details. The intensity of leg and back pain prior to PEA was assessed using a subjective visual analog scale (VAS) calibrated from 0 to 10 (0 = no pain and 10 = the worst pain imaginable). The patients' symptoms relief was rated using a Likert scale: 5 = greatly relief; 4 = some residual symptoms and symptoms relief > 50%; 3 = some residual symptoms and symptoms relief = 50%; 2 = residual symptoms and symptoms relief < 50%; 1 = no symptoms relief. For the comparison of clinical outcomes according to the symptoms relief, patients with grade 3, grade 4, and grade 5 were assigned to a group exhibiting >= 50% symptoms relief, while patients with grade 1 and grade 2 were assigned to a group exhibiting < 50% symptoms relief. Regarding the radiation exposure of PEA, simulations were performed with patient-speciﬁc input parameters (weight and length) and the actual 3D-RE system settings for each frame, including the automatic modulation of beam energy and dose level, and collimation. Effective dose (ED), which has been generally accepted single number index reﬂecting patient radiation risk, was subsequently calculated using the latest ICRP 103 weighing factors, published in 2007 [14].

StatisticalAnalysis. Age, the duration of discomfort prior to PEA, and VAS scores are expressed as means ±standard deviations. Demographic data within the two groups of greater symptoms relief and less were compared by using the chi-square test or the Fisher's exact test or unpaired t-test. Inter-reader agreement was evaluated using the intra-class correlation coefficients (ICCs), calculated according to Landis and Koch[15], for the contrast distribution of CE and 3D-RE. Simple linear regression analysis was used to determine the prediction of the outcome of PEA by the contrast distribution of CE and 3D-RE. All statistical analyses were performed using the Statistical Package for the Social Sciences software (SPSS Inc., Chicago, Illinois, USA). A P value of <0.05 was considered statistically signiﬁcant.

ELIGIBILITY:
Inclusion Criteria:

* FBSS or SS with unilateral radiculopathy.
* History of discogenic or radicular symptoms refractory to conservative treatments and epidural steroid injection for a minimum of 6 weeks.
* The PEA was standardized to all patients receiving the procedure.
* Each patient received an epidural injection, and if the symptoms persisted or the relief was insufficient, the patient received PEA >6-week interval between the epidural steroid injection.
* Positive provocative test during PEA was used to confirm the affected spinal level.
* All patients underwent CE before and after PEA; and 3D-RE after PEA.

Exclusion Criteria:

* History of spinal surgery and those with cauda equina syndrome
* Bleeding diathesis
* Associated somatic or psychiatric disease
* Vertebral fractures
* Pregnancy
* Tumors
* Other underlying systemic diseases that could signiﬁcantly influence the procedural outcomes were excluded.
* Bilateral symptoms
* Did not react to the provocation during PEA

Max Age: 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients who had FBSS or SS with unilateral radiculopathy underwent PEA.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Symptoms change after PEA | 1 month
  For the comparison of clinical outcomes according to the symptoms change, the participants' symptoms change was rated using a Likert scale to defined two groups by exhibiting >= 50% symptoms change and < 50% symptoms change.
Reproducibility of CE and 3D-RE | 1 month
  Inter-reader agreement was evaluated using the intra-class correlation coefficients (ICCs), calculated according to Landis and Koch, for the contrast distribution of CE and 3D-RE.
Usefulness of 3D-RE for predicting the outcome of PEA | 3 months
  Simple linear regression analysis was used to determine the prediction of the outcome of PEA by the contrast distribution of CE and 3D-RE.

SECONDARY OUTCOMES:
Radiation exposure of PEA | 1 month
  Regarding the radiation exposure of PEA, simulations were performed with patient-speciﬁc input parameters (weight and length) and the actual 3D-RE system settings for each frame, including the automatic modulation of beam energy and dose level, and collimation. Effective dose (ED), which has been generally accepted single number index reﬂecting patient radiation risk, was subsequently calculated using the latest ICRP 103 weighing factors, published in 2007.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chih Hsu, M.D., Study Director — Department of Radiology Tri-Service General Hospital National Defense Medical Center
Locations (1):
- No. 325, Sec. 2, Cheng-kung Rd., Neihu 114, Taipei, Taiwan, R.o.c., Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Manchikanti L, Helm Ii S, Pampati V, Racz GB. Percutaneous adhesiolysis procedures in the medicare population: analysis of utilization and growth patterns from 2000 to 2011. Pain Physician. 2014 Mar-Apr;17(2):E129-39. PMID 24658484
- [Background] Gerdesmeyer L, Wagenpfeil S, Birkenmaier C, Veihelmann A, Hauschild M, Wagner K, Muderis MA, Gollwitzer H, Diehl P, Toepfer A. Percutaneous epidural lysis of adhesions in chronic lumbar radicular pain: a randomized, double-blind, placebo-controlled trial. Pain Physician. 2013 May-Jun;16(3):185-96. PMID 23703406
- [Background] Racz GB, Heavner JE, Trescot A. Percutaneous lysis of epidural adhesions--evidence for safety and efficacy. Pain Pract. 2008 Jul-Aug;8(4):277-86. doi: 10.1111/j.1533-2500.2008.00203.x. Epub 2008 May 23. PMID 18503627
- [Background] Park SH, Ji GY, Cho PG, Shin DA, Yoon YS, Kim KN, Oh CH. Clinical Significance of Epidurography Contrast Patterns after Adhesiolysis during Lumbar Percutaneous Epidural Neuroplasty. Pain Res Manag. 2018 Apr 1;2018:6268045. doi: 10.1155/2018/6268045. eCollection 2018. PMID 29808106
- [Background] Kim JH, Jung HJ, Nahm FS, Lee PB. Does improvement in epidurography following percutaneous epidural neuroplasty correspond to patient outcome? Pain Pract. 2015 Jun;15(5):407-13. doi: 10.1111/papr.12197. Epub 2014 Apr 21. PMID 24750546
- [Background] Gupta R, Singh S, Kaur S, Singh K, Aujla K. Correlation between Epidurographic Contrast Flow Patterns and Clinical Effectiveness in Chronic Lumbar Discogenic Radicular Pain Treated with Epidural Steroid Injections Via Different Approaches. Korean J Pain. 2014 Oct;27(4):353-9. doi: 10.3344/kjp.2014.27.4.353. Epub 2014 Oct 1. PMID 25317285
- [Background] Hong Park C, Ho Lee S. Epidurographic Findings Following Percutaneous Epidural Adhesiolysis Failed to Correlate with Level of Pain Reduction in Patients with Lumbar Spinal Stenosis. Pain Med. 2017 May 1;18(5):842-845. doi: 10.1093/pm/pnw244. PMID 27651508
- [Background] Shin JW. Is epidurogram a reliable tool for the diagnosis of epidural adhesion? Korean J Pain. 2012 Apr;25(2):133-4. doi: 10.3344/kjp.2012.25.2.133. Epub 2012 Apr 4. No abstract available. PMID 22514786
- [Background] Kufeld M, Claus B, Campi A, Lanksch WR, Benndorf G. Three-dimensional rotational myelography. AJNR Am J Neuroradiol. 2003 Aug;24(7):1290-3. PMID 12917114
- [Background] El-Sheik M, Heverhagen JT, Alfke H, Froelich JJ, Hornegger J, Brunner T, Klose KJ, Wagner HJ. Multiplanar reconstructions and three-dimensional imaging (computed rotational osteography) of complex fractures by using a C-arm system: initial results. Radiology. 2001 Dec;221(3):843-9. doi: 10.1148/radiol.2213010606. PMID 11719688
- [Background] Manchikanti L, Boswell MV, Rivera JJ, Pampati VS, Damron KS, McManus CD, Brandon DE, Wilson SR. [ISRCTN 16558617] A randomized, controlled trial of spinal endoscopic adhesiolysis in chronic refractory low back and lower extremity pain. BMC Anesthesiol. 2005 Jul 6;5:10. doi: 10.1186/1471-2253-5-10. PMID 16000173
- [Background] Moon SH, Lee JI, Cho HS, Shin JW, Koh WU. Factors for Predicting Favorable Outcome of Percutaneous Epidural Adhesiolysis for Lumbar Disc Herniation. Pain Res Manag. 2017;2017:1494538. doi: 10.1155/2017/1494538. Epub 2017 Jan 26. PMID 28246488
- [Background] Wiesent K, Barth K, Navab N, Durlak P, Brunner T, Schuetz O, Seissler W. Enhanced 3-D-reconstruction algorithm for C-arm systems suitable for interventional procedures. IEEE Trans Med Imaging. 2000 May;19(5):391-403. doi: 10.1109/42.870250. PMID 11021683
- [Background] The 2007 Recommendations of the International Commission on Radiological Protection. ICRP publication 103. Ann ICRP. 2007;37(2-4):1-332. doi: 10.1016/j.icrp.2007.10.003. PMID 18082557